CLINICAL TRIAL: NCT01491581
Title: Efficacy of a Milk-based Nutrient-rich Bar on Nutritional Status and Cognitive Performance of School Children in Vietnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Can Tho University (Other); National Institute of Nutrition, Vietnam (Other Government); Global Alliance for Improved Nutrition (Other); ILSI, Japan (Unknown)
Responsible Party: Principal Investigator, Frank Wieringa, Senior Researcher, Institut de Recherche pour le Developpement
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: VietnamSchoolBar_2011
Record Dates: First submitted 2011-11-28; First posted 2011-12-14 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Cognitive Performance
Keywords: anthropometry; zinc; iodine; vitamin D; calcium; school children; food supplement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- micronutrient enriched bar (Experimental): bar enriched with micronutrients
  Interventions: Dietary Supplement: food bar
- control arm (Placebo Comparator): normal bar
  Interventions: Dietary Supplement: food bar

INTERVENTIONS:
Dietary Supplement: food bar — milk based food bar enriched with micronutrients
  Other Names: Goody

SUMMARY:
The objective of the study is to evaluate the impact of the milk-based nutrient-rich bar, specifically the effect of its fortification with zinc, iodine, vitamins A and D and calcium on nutritional status of school children, focusing on vitamin A and, zinc, iodine, calcium and iron status, and on their cognitive performances.

DETAILED DESCRIPTION:
Design: double-masked randomized control trial Place: three schools in South Vietnam, Can Tho district, South Vietnam Subjects: School children aged 6 to 10 years old, from first grade to third grade of 3 primary schools.

Duration of intervention: 6 months (consumption of Goody or "control bar")

Study groups: 2 groups:

Group 1: children will receive micronutrient enriched milk bar. Group 2: children will receive the same milk-based food except for the micronutrient fortification.

ELIGIBILITY:
Inclusion Criteria:

* pupil in one of the 2 selected schools, in grade 1 - 3
* weight for height > -3 z-scores
* hemoglobin concentration > 70 g/L

Exclusion Criteria:

* weight for height < -3 z-scores
* hemoglobin concentration <= 70 g/L

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 415 (Actual)
Dates: Start 2011-12; Primary Completion 2012-05 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
micronutrient status | 6 months intervention study with baseline and endpoint data collection
  change in micronutrient status (hemoglobin and serum concentrations of vitamin D, calium, zinc) from baseline to end of the intervention when children have received the food bar for 6 months, 5 days/week.

SECONDARY OUTCOMES:
cognitive function | 6 months intervention study with baseline and endpoint data collection
  change in cognitive function (as measured by Raven's test) in children from baseline to end point, when the children have received 6 months of food bar, 5 days/week

CONTACTS AND LOCATIONS:
Locations (1):
- Can Do primary school, Can Do, Can Tho City, Vietnam